CLINICAL TRIAL: NCT00151541
Title: A Phase 3, Randomized, Double-blind, Multi-dose Study to Evaluate the Safety and Efficacy of 5% Dapsone Topical Gel, (DTG 5%) When Co-administered With Vehicle Control, Adapalene Gel 0.1% or Benzoyl Peroxide Gel 4% in the Treatment of Acne Vulgaris.
Brief Title: A Phase 3 Study to Compare the Safety and Efficacy of 5% Dapsone Topical Gel, (DTG) Twice Daily in Combination With Once Daily Vehicle Control, Adapalene Gel 0.1% or Benzoyl Peroxide Gel 4%
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAP0407
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris; Acne; Dermatology; Dapsone; Dapsone Topical Gel
MeSH Terms: conditions — Acne Vulgaris

INTERVENTIONS:
Drug: Dapsone Topical Gel + adapalene gel 0.1%
Drug: Dapsone Topical Gel + benzoyl peroxide gel 4%
Drug: Dapsone Topical Gel + vehicle control

SUMMARY:
The purpose of this study is to compare the safety and efficacy of 5% Dapsone Topical Gel, (DTG) twice daily in combination with once daily vehicle control, adapalene gel 0.1% or benzoyl peroxide gel 4%. The second objective of the study is to determine dapsone exposure after co-administration of DTG 5% with vehicle control, adapalene or benzoyl peroxide gel.

DETAILED DESCRIPTION:
This is a 3 arm, 12-week, randomized, double-blind, multicenter study comparing safety and efficacy of DTG 5% twice daily plus vehicle control once daily vs. DTG 5% twice daily plus adapalene gel 0.1% once daily vs. DTG 5% twice daily plus 4% benzoyl peroxide gel once daily in subjects with acne vulgaris. Approximately 300 male and female subjects, 12 years of age and older, with acne vulgaris and > 20 inflammatory lesions (papules and/or pustules) and > 20 non-inflammatory lesions (comedones) above the mandibular line at Baseline will be enrolled. Follow-up visits will occur at Week 2, 4, 8 and 12. Global Acne Assessments, Lesion Counts and Local Adverse Reaction Assessments will be conducted at each visit. A physical exam will be done at Baseline and Week 12. Plasma Dapsone Level samples will be drawn at Baseline, Week 2 and Week 12/ET for dapsone plasma level assessments. Adverse events and concomitant medications will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

Study subjects will be considered for participation based upon medical history and findings from the pre-study interview and examination. They will be enrolled according to the following conditions:

1. Each subject or parent/guardian will read and sign the informed assent and/or consent form as required by IRB regulations. If a subject should require someone to read and/or interpret any or all of the informed consent, a statement of this fact will be documented. If a subject is unable to read or if a legally acceptable representative is unable to read, an impartial witness should be present during the entire informed consent discussion to ensure accurate representation of the informed consent document is given verbally. If a subject does not understand English, a validated translated informed consent agreement will be provided. If the subject is a minor, the signature of their parent or guardian will be required per Institutional Review Board regulations.
2. Male and female subjects, 12 years of age and older.
3. A female subject of childbearing potential must not be pregnant or nursing. All female subjects must be practicing an effective method of birth control as determined by the Investigator. Any female who is not sexually active must agree to begin using an effective method of birth control, excluding hormonal birth control, if she becomes sexually active during the study.

   A female subject using hormonal birth control must have been on a stable dose for 3 months prior to Baseline.

   Note: A surgically sterilized partner is not an acceptable method of birth control.
4. A urine pregnancy test will be required of all female subjects, 60 years of age and younger prior to treatment. If the subject can provide documentation of surgical sterilization, at the baseline visit, a pregnancy test is not required.

   Negative test results must be obtained prior to randomization.
5. Subjects must be in good physical and mental health.
6. The subject must be willing to avoid swimming and bathing for 2 hours following test article application. Additionally, the subject must be willing to avoid moisturizers, sunscreens and cosmetics for 1 hour following test article application.
7. The subject must score > 2 on the Global Acne Assessment Score at Baseline (Appendix D).
8. Subjects must have a clear diagnosis of acne vulgaris of the face, and have a minimum of 20 inflammatory lesions (pustules and papules) and 20 non-inflammatory lesions (comedones) above the mandibular line at Baseline. If, in the judgment of the Investigator, the subject's acne should be treated with a systemic acne medication, they should not be enrolled in the study.
9. Subjects must be willing to undergo blood draws throughout the study.
10. The subject must be willing and able to comply with the requirements of the protocol

Exclusion Criteria:

MEDICATIONS EXCLUDED IN THE ADMISSION CRITERIA WILL NOT BE PERMITTED DURING THE STUDY.

Subjects who meet any of the following criteria will be excluded from study entry:

1. Subjects using systemic immunosuppressive medications within 28 days prior to Baseline and throughout the study. Intranasal and/or inhaled corticosteriods are acceptable throughout the study if at a stable and standard dose, as labeled within the Package Insert.
2. Subjects who are using topical agents for acne (including and not limited to benzoyl peroxide, antibiotics, topical vitamin A derivates such as retinol or retinoids, medicated cosmetics, cleansers) within 14 days prior to Baseline and throughout the study. This includes over the counter medications and cleansers that contain acne treatment ingredients, e.g. benzoyl peroxide, salicylic acid.
3. Subjects who have received light therapies (ultraviolet B, tanning bed, lasers, photodynamic treatment), systemic medications, or skin treatments known to affect acne or inflammatory responses within the 28 days prior to Baseline and throughout the study. This includes but is not limited to: antibiotics, large doses (>50,000 U/day) of vitamin A, hormones (excluding those used for birth control), spironolactone, aldactone, aldactizide, cyproterone acetate, NSAIDS and chemical exfoliative treatments (alpha-hydroxy acid or "fruit-wash," "lunchtime" or phenol peels) or physical peels (laser, "dry ice" peels). Short-term treatment with antibiotics and NSAIDS during the study for non-acne related conditions is acceptable provided that exposure is limited to 14 days per course for antibiotics and 7 days per month for NSAIDS.
4. Subjects who have received isotretinoin (Accutane) within the three months prior to Baseline and throughout the study.
5. Subjects that have participated in any previous QLT USA, Inc. (formerly Atrix Laboratories, Inc.) dapsone topical gel studies.
6. Subjects who have any medical condition which, in the Investigator's judgment, makes the subject an inappropriate study candidate.
7. Subjects who have any condition that would hinder accurate facial acne evaluations including excessive facial hair (beard), excessive scarring, sunburn or other disfigurement.
8. Subjects with severe cystic acne or acne conglobata.
9. Subjects with any active or developing nodules above the mandibular line at Baseline.
10. Subjects with a known allergy or hypersensitivity to dapsone, adapalene, benzoyl peroxide, or any component of the study products.
11. Subjects taking another investigational test article within the 30 days prior to Baseline or throughout the study.
12. Female subjects having started a new, or having changed their current hormonal contraceptive or hormone replacement therapy within three months prior to Baseline. Subjects receiving Depo Provera® injections in preceding 4 months are excluded from the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2005-02; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint will be mean percent reduction in inflammatory lesion counts.

SECONDARY OUTCOMES:
Additional efficacy endpoints will be the mean percent reduction from Baseline in non-inflammatory and total lesion counts, as well as the proportion of subjects who achieve success (none/minimal) on a 5-point Global Acne Assessment Score.
Safety endpoints will include treatment-emergent and treatment related adverse events. An additional safety endpoint will be the local adverse reaction assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Garrett, MS, DDS, FACS, Study Director — QLT USA, Inc.